CLINICAL TRIAL: NCT06647667
Title: High Interval Versus Moderate Intensity Continuous Training on Soluble st2 Biomarkers in Chronic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Reda Ali, PhD candidate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P.T.REC/012/004017
Record Dates: First submitted 2024-06-14; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure
Keywords: sST2 biomarker; Minnesota Questionare; HIITS
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: 1. Patients will receive high intensity interval training (HIIT)
  2. Patients will receive moderate intensity continuous training (MICT)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): high intensity interval training
  Interventions: Other: HIITS
- group B (Experimental): moderate intensity continuous training
  Interventions: Other: MICT

INTERVENTIONS:
Other: HIITS — Frequency: HIIT will be in 2 supervised sessions per week for 12 weeks on the treadmill.
  session duration from 30-40 min including the waming up and cooling down Intensity: HIIT included 4 minute intervals aiming 60-85% of heart rate reserve
  Arms: group A
Other: MICT — Frequency: Moderate continuous training is scheduled 2 times per week for 12 weeks.
  Intensity: exercise had been applied on the treadmill with 40%-59% of heart rate reserve) session duration from 30-40 min including the warming up and cooling down
  Arms: group B

SUMMARY:
This study was designed to compare between the effect of high intensity interval training (HIIT) and moderate intensity continuous training (MICT) on soluble ST2 biomarkers among chronic heart failure patients, also measure the improvement in the quality of life with different modes of exercise and with of it is more benifitial for the heart failure patient

DETAILED DESCRIPTION:
The data concerned with the study including soluble ST2 biomarker levels, ejection fraction and MLHFQ was measured before and after twelve weeks of treatment.In this study a total sixty male patients with chronic heart failure NYHA class (I &II) were selected from the outpatient clinic, El-Demerdash hospital, Ain-shams University. Their age ranged from 50-60 years. Patients were randomly assigned into two groups, group A receiving HIIT along with prescribed medical treatment and group B receiving MCT along with prescribed medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* The patients selection was according to the following criteria:

  * Patients diagnosed with chronic heart failure (New York heart association class I& II) with systolic left ventricular dysfunction.
  * Their left ventricular ejection fraction (LVEF) <40%.
  * Medical treatment was optimized at least three months prior to study entry.
  * All patients didn't participate in any rehabilitation programs prior to the study.

Exclusion Criteria:

* Patients who had met one of the following criteria were excluded from the study:

  1. Signs of acute heart failure, unstable angina or severe arrhythmia three months prior to enrolment in the study.
  2. Pacemakers.
  3. Chronic obstructive pulmonary disease.
  4. Other disorders counteracting exercise testing conditions that limit lower limb mobility (for example, burns, fractures)
  5. Pre-existing neuromuscular diseases (for example Myasthenia Gravis).

Ages: 50 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
soluble ST2 biomarker level | before the start of the trail and at the end of the trail 3 months
  sample was taken at the cubited vein at the beginning of the program and also at its end

SECONDARY OUTCOMES:
ejection fraction | before the start of the trail and at the end of the trail 3 months
  Left ventricular systolic dysfunction was assessed using the ejection fraction by 2D simpson method
mannisota of daily living questionnaire score | before the start of the trail and at the end of the trail 3 months
  The twenty one item questionnaire was usedfrom 0 (none) to 5 (very much). It provides a total score (range 0-105, from best to worst HRQoL), as well as scores for two dimensions, physical (8 items, range 0-40) and emotional (5 items, range 0-25). The other eight items (of the total of 21) are only considered for the calculation of the total score.
peak exercise response | before the start of the trail and at the end of the trail 3 months
  monitoring the peak exercise response

CONTACTS AND LOCATIONS:
Overall Officials: Donia M Elmasry, Doctorate, Study Director — Cairo University
Locations (1):
- Faculty of physical therapy Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
study protocol and final results
Supporting Information: Study Protocol, ICF
Time Frame: August 2024 till December 2024
Access Criteria: researchers

DOCUMENTS (1):
  • Study Protocol (2022-09-11): https://cdn.clinicaltrials.gov/large-docs/67/NCT06647667/Prot_000.pdf